CLINICAL TRIAL: NCT07253116
Title: A Phase I/II, Dose-Escalation, Dose-Expansion, and Efficacy-Expansion Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Preliminary Efficacy of WJ22096 Tablets Administered Orally in Patients With Advanced Solid Tumors
Brief Title: A Phase I/II Clinical Study of WJ22096 Tablets in Patients With Advanced Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Nanjing Jingao biomidical technology Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: WJ22096-001-I
Record Dates: First submitted 2025-11-19; First posted 2025-11-28 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Advanced Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental：WJ22096 tablets (Experimental): WJ22096 orally once daily after meal
  Interventions: Drug: WJ22096

INTERVENTIONS:
Drug: WJ22096 — WJ22096: orally once daily after meal

SUMMARY:
This is a Phase I/II, open-label, preliminary study of safety, tolerability, pharmacokinetics, and efficacy. The study comprises three parts: a Dose Escalation cohort, a Dose Expansion cohort, and an Efficacy Expansion cohort.

Dose Escalation cohort aims to evaluate the safety, tolerability, pharmacokinetic (PK) characteristics, and preliminary efficacy of WJ22096 Tablets in patients with advanced solid tumors for whom standard therapies have failed, are not tolerated, or for whom no standard therapy exists.

Dose Expansion cohort Based on an evaluation of preliminary data, the Sponsor and the Safety Monitoring Committee (SMC) will select 1-2 dose levels to further evaluate preliminary efficacy, safety, tolerability, and PK characteristics, and to confirm the Recommended Phase 2 Dose (RP2D). Each dose cohort will enroll approximately 9-12 subjects with advanced solid tumors (for whom standard therapies have failed, are not tolerated, or for whom no standard therapy exists), predominantly comprising patients with Non-Small Cell Lung Cancer (NSCLC), Colorectal Cancer (CRC), and Pancreatic Cancer.

Efficacy Expansion cohort aims to evaluate the efficacy, safety, tolerability, and PK characteristics at the selected dose in patients with specific tumor types, such as NSCLC, CRC, and Pancreatic Cancer. The dosing regimen will be the RP2D determined during the Dose Escalation and Dose Expansion cohorts. It is initially planned to expand 2-3 cohorts using Simon's two-stage minimax design, with approximately 20-40 subjects planned for enrollment in each cohort. (The specific tumor types for expansion, sample size, and number of cohorts will be adjusted by the Principal Investigator (PI) and the Sponsor based on results from the preceding stages of the trial).

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary participation in this study, with a signed informed consent form (ICF) provided after being fully informed;
2. Age ≥ 18 years, regardless of sex;
3. Histologically and/or cytologically confirmed diagnosis of advanced solid tumors, who have failed standard therapy, are intolerant to standard therapy, or for whom no standard therapy is available;
4. Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1;
5. Estimated life expectancy > 12 weeks;
6. Adequate hematological and organ function, with the following laboratory results obtained within 7 days prior to the first administration of the study drug (no blood transfusions, hematopoietic stimulating factors, or human albumin preparations within 14 days prior to the test):

   * Absolute neutrophil count (ANC) ≥ 1.5 x 10⁹/L
   * Platelets (PLT) ≥ 100 x 10⁹/L
   * Hemoglobin (Hb) > 90 g/L
   * Aspartate aminotransferase (AST) and Alanine aminotransferase (ALT) ≤ 3.0 × upper limit of normal (ULN) (or ≤ 5 × ULN if liver metastases are present);
   * Total bilirubin ≤1.5 × ULN;
   * Serum creatinine ≤ 1.5 × ULN or creatinine clearance (Ccr, calculated using the Cockcroft-Gault formula) ≥ 45 mL/min;
7. All acute toxicities from prior anti-tumor therapies or surgical procedures must have resolved to baseline severity or to ≤ Grade 1 according to NCI CTCAE v5.0 (exceptions include alopecia or pigmentation);
8. Female subjects of childbearing potential (WOCBP) must have a negative serum pregnancy test within 7 days prior to the first dose and agree to use effective contraceptive measures during the study drug administration period and for 3 months after the last dose. Male subjects whose sexual partners are WOCBP must agree to use effective contraceptive measures during the study drug administration period and for 3 months after the last dose.

   Specific Inclusion Criteria:
9. At least one measurable tumor lesion as defined by RECIST v1.1, with no biopsy of the target lesion within the prior 2 weeks (Applicable to dose expansion and efficacy expansion cohorts);
10. The Non-Small Cell Lung Cancer (NSCLC) cohort will prioritize the enrollment of subjects with G12C mutations (Applicable to the efficacy expansion cohort);
11. Subjects with pancreatic cancer must have received ≤2 prior lines of therapy (Applicable to dose expansion and efficacy expansion cohort).

Exclusion Criteria:

1. General Conditions 1) Pregnant or lactating women; 2) Known allergy or contraindication to any components of the study drug; 3) History of drug abuse; 4) History of alcohol abuse (alcoholism); 5) Difficulty with intravenous blood collection (e.g., history of needle phobia, hemophobia).
2. Prior or Concomitant Therapies 1) Prior or current treatment with a FAK inhibitor; 2) Received systemic anti-tumor drug therapy (e.g., chemotherapy, targeted therapy, endocrine therapy) within 3 weeks prior to the first dose (or, if prior anti-tumor drug therapy was received, a washout period of 5 half-lives, whichever is longer), or radiotherapy within 3 weeks, or immunotherapy within 4 weeks prior to the first dose; 3) Use of Chinese herbal medicine with anti-tumor effects within 2 weeks prior to the first dose; 4) Concomitant use of moderate or strong inhibitors or inducers of CYP3A, or other products (e.g., grapefruit juice), or inhibitors or inducers of P-gp; or discontinuation of such agents for less than 5 half-lives or 14 days (whichever is longer) prior to the first dose; 5) Known history of organ transplant or stem cell transplant; major surgery within 4 weeks prior to the first dose, or planned surgery during the study period; 6) Radiotherapy within 21 days prior to administration (Exception: Patients who received radiotherapy to ≤5% of their bone marrow volume are eligible regardless of when the radiotherapy was received).
3. Medical History, Current Conditions, and Laboratory Abnormalities 1) Active gastrointestinal (GI) abnormalities including, but not limited to: inability to take oral medication, requirement for IV nutritional support, peptic ulcers, chronic diarrhea (e.g., Crohn's disease, irritable bowel syndrome), or vomiting, or other factors that, in the investigator's opinion, may significantly affect drug absorption, metabolism, or excretion (e.g., small bowel stom); 2) Clinically uncontrolled third-space fluid accumulation, such as pleural effusion, pericardial effusion, ascites, or pelvic effusion, deemed unsuitable for enrollment by the Investigator; 3) Patients with active brain metastases, including symptomatic brain metastases, meningeal metastases, or spinal cord compression. However, the following patients are allowed: a. Patients with treated brain metastases (e.g., surgery, radiotherapy) who are radiologically stable for at least 4 weeks prior to the first dose, and/or have no new or progressive neurological symptoms or signs, no evidence of new or enlarging brain metastases, and have discontinued systemic corticosteroid therapy (dose >10 mg/day prednisone or equivalent) for at least 4 weeks prior to the first dose; b. Subjects with untreated, asymptomatic brain metastases who do not require corticosteroids; 4) Poorly controlled hypertension: systolic blood pressure ≥160 mmHg and/or diastolic blood pressure ≥100 mmHg during the screening period; 5) Uncontrolled diabetes mellitus (baseline fasting blood glucose >8.9 mmol/L or Glycosylated Hemoglobin (HbA1c) >6.5%); 6) Clinically significant bleeding symptoms or obvious bleeding tendency within 4 weeks prior to the first dose (e.g., gastrointestinal bleeding, peptic ulcer bleeding); 7) Active HBV or HCV infection: If HBsAg is positive or/and anti-HBc is positive, HBV DNA must be tested to confirm it is above the limit of quantitation; If anti-HCV is positive, HCV RNA must be tested to confirm HCV viral load is above the limit of quantitation; 8) Human Immunodeficiency Virus (HIV) infection or a known history of positive HIV serology; 9) History of syphilis with positive results for both specific (treponemal) and non-specific (non-treponemal) syphilis antibodies; 10) Presence of concurrent malignancies within 5 years prior to enrollment (Exceptions: adequately treated cervical carcinoma in situ, non-melanoma skin cancer or lentigo maligna, localized cutaneous squamous cell carcinoma, basal cell carcinoma, prostate cancer not requiring anti-tumor treatment, thyroid cancer, ductal carcinoma in situ of the breast, and urothelial carcinoma ≤T1); 11) Occurrence within 6 months prior to the first dose of: acute coronary syndrome, congestive heart failure (New York Heart Association [NYHA] functional class ≥II), left ventricular ejection fraction (LVEF) <50%, cerebrovascular accident, transient ischemic attack, stroke, deep vein thrombosis, pulmonary embolism, aneurysm, arterial dissection, or other Grade 3 or higher cardiovascular or cerebrovascular events; 12) Arrhythmias (e.g., bradyarrhythmias) or conduction abnormalities considered clinically significant by the Investigator, congenital long QT syndrome, or unmeasurable or Fridericia's-corrected QTc >450 ms for males or >470 ms for females; 13) Presence of persistent or severe active infectious diseases (including bacterial, fungal, viral, etc.) requiring intravenous anti-infective therapy; 14) Known or suspected refractory urinary tract infection (UTI) or a history of recurrent UTIs (≥3 episodes in the past 12 months); 15) Any other condition that, in the opinion of the investigator, may affect study results or interfere with full participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-11-20 (Actual); Primary Completion 2028-11-30 (Estimated); Study Completion 2028-11-30 (Estimated)

PRIMARY OUTCOMES:
DLT (Dose Limiting Toxicity) | up to 3 years
  It is suitable for dose escalation .DLT is defined as any of AE that Safety Monitoring Committee considers to have occurred during the DLT observation period and may be causally related to WJ22096 and meet DLTcriteria.
Adverse Events (AE) / Serious Adverse Events (SAE) | up to 3 years
  Incidence and severity of adverse events (AE) and serious adverse events (SAE) as assessed according to NCI-CTCAE 5.0, as well as abnormalities in physical examination, ECOG score, vital signs, electrocardiogram, ophthalmic tests and laboratory tests.
MTD (Maximal Tolerable Dose) | up to 3 years
  Defined as the dose level at which the estimated toxicity probability is closest to the target toxicity probability during the DLT observation period
RP2D (Recommended Phase 2 Dose) | up to 3 years
  RP2D will be determined based on a combination of safety, tolerability, PK and/or pharmacodynamic studies .
ORR (Objective Response Rate) (efficacy expansion cohort) | up to 3 years
  It is suitable for the curative effect development stage.Objective Response Rate by RECIST 1.1.

SECONDARY OUTCOMES:
Cmax | up to 3 years
  Maximum Plasma Concentration
Tmax | up to 3 years
  Time to Cmax
AUC0-t | up to 3 years
  Area under the concentration versus time curve from time 0 to the last measurable concentration
AUC0-inf | up to 3 years
  AUC from time 0 to infinity
t1/2 | up to 3 years
  Elimination half life time
CL/F | up to 3 years
  Apparent Clearance
Vd/F | up to 3 years
  Apparent volume of distribution
RAC | up to 3 years
  Accumulation index
FD | up to 3 years
  degree of fluctuation
DOR | up to 3 years
  Duration of response
DCR | up to 3 years
  Disease Control Rate
PFS | up to 3 years
  Progression-free survival
OS | up to 3 years
  Overall survival
ORR (dose escalation and dose expansion stage) | up to 3 years
  It is suitable for the curative effect development stage.Objective Response Rate by RECIST 1.1.
adverse events (AE) and serious adverse events (SAE) (efficacy expansion stage) | up to 3 years
  To evaluate incidence, severity and outcome of adverse events (AE),and serious adverse events (SAE)

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided